CLINICAL TRIAL: NCT06916286
Title: A Prospective, Randomized, Multi-center Trial Evaluating the Effect of Surgical Drain Securement on Patient Quality of Life and Postoperative Drain-related Complications
Brief Title: Evaluating the Effect of Surgical Drain Securement on Patient Quality of Life and Postoperative Drain-related Complications
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: University of Mississippi Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00128120
Record Dates: First submitted 2025-03-31; First posted 2025-04-08 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-03

CONDITIONS: Surgical Drain
Keywords: Drain Insertion Site; Drain Site Complication; Plastic and Reconstructive Surgery
MeSH Terms: interventions — Sutures

STUDY DESIGN:
Intervention Model Description: On the day of surgery, patients will be randomized to either A) drains being secured with the K-Lock device or B) drains being secured with the suture-based technique. All drains will be secured according to randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- K-Lock Device (Experimental): K-Lock securement device
  Interventions: Device: K-Lock
- Traditional Suture (Active Comparator): Traditional suture securement
  Interventions: Other: Suture

INTERVENTIONS:
Device: K-Lock — Surgical drain securement with a novel sutureless K-LOCK device
  Arms: K-Lock Device
Other: Suture — Surgical drain securement with traditional suture-based methods
  Arms: Traditional Suture

SUMMARY:
The objective of this study is to evaluate whether surgical drain securement with a novel sutureless device (K-LOCKTM) will improve patient quality of life and reduce postoperative drain-related complications compared to drain securement with traditional suture-based methods. The K-LOCK™ Device is a novel sutureless drain securement device that may improve patient experiences with surgical drains.

DETAILED DESCRIPTION:
Patients will be identified as potential subjects where the study team will speak with them, determine eligibility, and obtain consent prior to surgery. On the day of surgery, patients will be randomized to either A) drains being secured with the K-Lock device or B) drains being secured with the suture-based technique. All drains will be secured according to randomization.

Postoperatively: The study team will follow the subjects weekly via the electronic medical record documenting (in REDCap) calls made to the triage nurse, visits to the emergency department, requests for additional pain medications, unexpected drain removal, need for additional drain placement, etc. Subjects will return to clinic at their regularly scheduled follow-up appointments with no additional study related activities and will be followed by the study team weekly, via chart review for a total of 3 months from their surgery date. When the subjects return to clinic to have their final drain removed they will be asked to complete a survey asking about their experience with their drains and drain securement. We will also have a blinded evaluator complete a short survey evaluating the skin around the drain insertion site. Photos will be taken of the drain site upon drain removal and again at the 3 month follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Patient of the Department of Plastic and Reconstructive Surgery
* Able to sign English language Consent form
* Undergoing a surgical procedure where placement of one or more surgical drains is anticipated

Exclusion Criteria:

* Unable to sign English language consent form
* Incompatible drain size placed
* Allergy or sensitivity to skin adhesives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Patient-Reported Outcome Measure Score | Month 3
  Patient reported outcome measures questionnaire will be completed by participant. Total score ranges from 6-30 with a higher score indicating a higher level of patient satisfaction.

SECONDARY OUTCOMES:
Number of Complications | Month 3
  Number of complications including calls to triage nurse, visits to Emergency Room, requests for additional pain medication, early loss of drain.
Rating of Drain Exit Sites | Month 3
  Questionnaire to be completed by a health care team member who is blinded to drain securement method. Drain site will be inspected for erythema, irritation, blistering, maceration, etc. and rated after removal of the drain. Ratings will range from 0-4 with higher rating indicating more severity.

CONTACTS AND LOCATIONS:
Overall Officials: Bennett W Calder, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No